CLINICAL TRIAL: NCT00839592
Title: Acupuncture Treatment of Primary Insomnia
Brief Title: Acupuncture for Primary Insomnia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Hong Kong Baptist University (Other); Hong Kong Professional Teachers' Union (Unknown)
Responsible Party: Dr. Chung Ka-Fai/ Associate Professor, the University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ACUP-001
Record Dates: First submitted 2009-02-06; First posted 2009-02-09 (Estimated); Last update posted 2010-01-14 (Estimated); Status verified 2010-01

CONDITIONS: Insomnia
Keywords: Insomnia; Acupuncture; Electroacupuncture; Randomized Clinical Trial; Traditional Chinese Medicine
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Electroacupuncture; Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Electroacupuncture (Experimental): Acupoints will be treated at bilateral Ear Shenmen, Sishencong (EX-HN1), Anmian, and unilateral Yintang (EX-HN3) and Baihui (GV20).
  Acupuncture will be performed by a registered Chinese medicine practitioner. "De qi"(an irradiating feeling considered to be indicative of effective needling) is achieved if possible. An electric-stimulator (CEFAR Acus II, Lund, Sweden) will be connected to these needles to give an electric-stimulation in continuous wave, frequency of 4 Hz, 0.45 ms square wave pulses and constant current. The needles will be left for 30 min and then removed. Acupuncture treatment will consist of three sessions per week for 3 consecutive weeks.
  Interventions: Other: Electroacupuncture
- Placebo Acupuncture (Placebo Comparator): Placebo needles designed by Streitberger (1998) will be used. The placebo needles are blunt needle that will not penetrate the skin during needle insertion. The handles of these placebo needles will slide over the needle when it is compressed, giving it the appearance of penetrating the skin. The placebo needles are inserted to the same acupoints as stated in the electroacupuncture group. The needles are held by a surgical tape or hair pin in hairy region to imitate the retention of needles. The needles are connected to an electric-stimulator with zero frequency and amplitude. The number, duration and frequency of the treatment sessions, and the intervention procedure will be the same for electro-acupuncture and placebo acupuncture.
  Interventions: Other: Electroacupuncture

INTERVENTIONS:
Other: Electroacupuncture — Acupuncture at bilateral Ear Shenmen, Sishencong EX-HN1, Anmian, and unilateral Yintang EX-HN3 and Baihui GV20. The needles will be left for 30 min and then removed. Acupuncture treatment will consist of three sessions per week for 3 consecutive weeks.
  Other Names: Acupuncture

SUMMARY:
This is a randomized controlled trial to evaluate acupuncture treatment on insomnia in the adult population in Hong Kong.

DETAILED DESCRIPTION:
Acupuncture is potential to be an alternative treatment for primary insomnia. The purpose of this study is to evaluate the clinical effectiveness of acupuncture treatment on primary insomnia. This is a randomized single-blinded controlled trial. Patients will be randomly assigned to the electro-acupuncture group or the placebo acupuncture group. Patients will be put into groups and then compared.

ELIGIBILITY:
Inclusion Criteria:

* Hong Kong residents
* aged 18-65
* Ethnic Chinese
* Meet the diagnosis criteria of primary insomnia for at least 3 months according to DSM-IV using the Structured Clinical Interview for DSM-IV (SCID)
* Willing to give informed consent
* total score of Insomnia Severity Index (ISI) at least 15
* Able to comply with trial protocol

Exclusion Criteria:

* Participation in any clinical trial during the previous 3 months prior to baseline
* Any current major depressive disorder, generalized anxiety disorders or panic disorder, manic or hypomanic episode, substance use disorders besides caffeine and nicotine, organic mental disorder, schizophrenia or any other psychotic disorder as defined by DSM-IV criteria
* Serious physical illness or mental disorders due to a general medical condition which is judged by the investigator to render unsafe
* Valvular heart defects, bleeding disorders or taking anticoagulant drugs.
* Any acupuncture treatment during the previous 12 months prior to baseline.
* In the investigator's opinion, the patient has a significant risk of suicide
* Pregnant, breast-feeding, or woman of childbearing potential not using adequate contraception
* Infection or abscess close to the site of selected acupoints and in the investigator's opinion inclusion is unsafe
* Herbal remedies, over-the-counter medications or psychotropic drugs, which are intended for insomnia, were taken within the last 2 weeks prior to baseline or during the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-07; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Self-rated sleep quality score measured by Insomnia Severity Index questionnaire | Baseline, weekly during the treatment course, 1-week posttreatment

SECONDARY OUTCOMES:
Sleep parameters (sleep onset latency, sleep efficiency, total sleep time, times of wakening during sleep) by objective measure - wrist actigraphy | Baseline, and 1-week posttreatment
Sleep parameters (sleep onset latency, sleep efficiency, total sleep time, times of wakening during sleep) by subjective measures using sleep log. | Baseline, weekly during the treatment course, and 1-week posttreatment
Self-rated sleep quality score measured by the Pittsburgh Sleep Quality Index (PSQI) questionnaire | Baseline, and 1-week posttreatment
Anxiety and depression states measured by Hospital Anxiety and Depression Scale (HADS) | Baseline, and 1-week posttreatment
Subjects' functioning regarding work/study, social life and family measured by Sheehan Disability Index | Baseline, and 1-week posttreatment
Subjects' credibility to the treatment measured by Credibility of treatment rating scale | Second and the last time of the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ka-Fai Chung, MBBS, Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

REFERENCES:
- [Derived] Yeung WF, Chung KF, Yu YB, Lao L. What predicts a positive response to acupuncture? A secondary analysis of three randomised controlled trials of insomnia. Acupunct Med. 2017 Mar;35(1):24-29. doi: 10.1136/acupmed-2016-011058. Epub 2016 Aug 8. PMID 27503746
- [Derived] Yeung WF, Chung KF, Zhang SP, Yap TG, Law AC. Electroacupuncture for primary insomnia: a randomized controlled trial. Sleep. 2009 Aug;32(8):1039-47. doi: 10.1093/sleep/32.8.1039. PMID 19725255